CLINICAL TRIAL: NCT03539120
Title: Prognosticating Outcomes in Stroke, Acquired Brain Injury, Amputee and Other Neurological Impairments
Brief Title: Post-amputation Survival Following Rehabilitation Medium and Long-term Follow up Study, a Retrospective Analysis.
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Shrikant Pande, senior consultant, Changi General Hospital
Other Study IDs: 201511-00072
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up for survival — No intervention, this is an observational study of survival outcomes.

SUMMARY:
This is a retrospective data analysis of patients who underwent lower limb amputation and rehabilitation and follow up.

Investigators analysed their survival outcomes in relation to various comorbidities i. e ischaemic heart disease, renal impairment, vascular interventions.

DETAILED DESCRIPTION:
Inclusion criteria: Patients admitted for major dysvascular lower limb amputation, with complete follow-up record available.

Exclusion criteria: Traumatic amputations, minor amputations, i.e. ray and toe amputation, and incomplete follow-up records.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted for major dysvascular lower limb amputation, with complete follow-up record available.

Exclusion criteria:

Exclusion Criteria:

Traumatic amputations, minor amputations, i.e. ray and toe amputation, and incomplete follow-up records

Age Groups: Child, Adult, Older Adult
Study Population: This study aimed to analyse survival outcome in patients with dysvascular lower limb amputation and identify relationship with existing comorbidities, i.e. diabetes mellitus (DM), peripheral vascular disease (PVD), ischaemic heart disease (IHD), estimated glomerular filtration rate (e-GFR), and chronic kidney disease (CKD). We also analysed the length of hospital stay, linear relationship with duration of DM, and vascular interventions.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
survival in relation to time | 6 months to 6 years
  Survival outcomes were analysed and have been included in the results.

IPD SHARING:
Plan to Share IPD: No